CLINICAL TRIAL: NCT05290610
Title: Intracranial Stimulation Mapping In Epilepsy -The InStim Study
Brief Title: Intracranial Stimulation Mapping In Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSYCH-2021-30271
Record Dates: First submitted 2022-01-21; First posted 2022-03-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Brain Mapping

STUDY DESIGN:
Intervention Model Description: This is a single group prospective feasibility study on adult epilepsy patients evaluating whether study tasks and workflow are feasible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Research IESM (Other): Functional mapping for research application
  Interventions: Other: Functional mapping

INTERVENTIONS:
Other: Functional mapping — Intracranial EEG data acquisition, observation and behavioral testing, and intracranial electrical stimulation

SUMMARY:
This is a single group prospective study to determine the feasibility for generating brain maps that localize cerebral functions and inter-regional information flow in partial epilepsy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years and older at screening.
* Written informed consent is obtained from the participant to comply with the requirements of the study.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Currently undergoing clinically indicated intracranial EEG monitoring for planning of epilepsy surgery in the University of Minnesota/MINCEP program.

Exclusion Criteria:

* Pregnancy ruled out prior to approval for intracranial EG monitoring.
* Persons who are rendered temporarily or permanently invulnerable by inability to understand the research due to study complexity, cognitive impairment, or by inability to make independent decisions owing to University of Minnesota or to Fairview health services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The effect of prefrontal direct electrical brain stimulation on cognitive effort | Immediately after stimulation sessions
  The change in subjective value of cognitive effort (area under the curve) after direct electrical brain stimulation to different areas of the prefrontal cortex during an effortful task

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Herman, MD, Principal Investigator — UMN
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05290610/ICF_000.pdf